CLINICAL TRIAL: NCT01167699
Title: An Open Study With OXN to Evaluate the Patient Preference for Pain Treatment With Respect to Quality of Life After WHO Stap I or Step II Analgesics for Patients With Moderate to Severe Non-malignant Pain
Brief Title: Oxycodone/Naloxone (OXN) Combination in Moderate to Severe Non-malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Pharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXN3501; 2008-001026-14 (EudraCT Number)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2011-07

CONDITIONS: Pain
Keywords: Oxycodone/naloxone; patient preference; WHO step I/II; Moderate to severe non-malignant pain
MeSH Terms: conditions — Pain; Patient Preference | interventions — Oxycodone; Naloxone

INTERVENTIONS:
Drug: Oxycodone and naloxone — Oxycodone hydrochloride and naloxone hydrochloride combination, prolonged release

SUMMARY:
The main objective of the study is to evaluate the patient preference for pain treatment with respect to quality of life in patients with moderate to severe non malignant pain. Patients who have insufficient pain relief and/or unacceptable side effects with the previous analgesic treatment WHO step 1 or 2 and require around-the-clock opioid therapy can be included in the study. The WHO step I or II analgesics will be compared with the new study medication OXN (oxycodone/naloxone).

DETAILED DESCRIPTION:
Patients will receive OXN for 3 weeks in the first phase (core phase) and in the second phase (extension phase) they will receive OXN as is daily clinical practice until reimbursement of OXN in the Netherlands or Belgium or until discontinuation on request of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years or older with moderate to severe non-malignant pain who are willing to provide written informed consent.
2. Females less than one year post-menopausal must have a negative urine pregnancy test recorded at the screening visit, be non-lactating, and willing to use adequate and reliable contraception throughout the study. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
3. Patients with documented history of moderate to severe, non-malignant pain treated with WHO step I or II analgesics with insufficient pain relief and/or unacceptable side effects that requires around-the-clock opioid therapy (starting dose of oxycodone over 20 mg/day) and are likely to benefit from WHO step III opioid therapy for the duration of the study. Patients must be willing to discontinue their current analgesics, like opioids. Co-analgesics, such as anti-depressants and anti-epileptics, can be continued provided that the co-analgesics are used on a stable dose before and during the study.
4. Patients are willing to discontinue pre study laxative medication.
5. Patients taking daily fibre supplementation or bulking agents are eligible if they can be maintained on a stable dose and regimen throughout the study, and in the investigators opinion are willing and able to maintain adequate hydration.
6. Patients willing and able to participate in all aspects of the study, including use of medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements as evidenced by providing written, informed consent.

Exclusion Criteria:

1. Any history of hypersensitivity to oxycodone, naloxone, related products, and other ingredients.
2. Patients that require a dose over 20 mg/day oxycodone at the start of the study.
3. Active alcohol or drug abuse and/or history of opioid abuse.
4. Evidence of clinically significant cardiovascular, renal, hepatic, or psychiatric disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination, that would place the patient at risk upon exposure to the study medication or that may confound the analysis and/or interpretation of the study results.
5. In the investigator's opinion, patients who are receiving hypnotics or other central nervous system (CNS) depressants that may pose a risk of additional CNS depression with opioid study medication.
6. Patients receiving opioid substitution therapy for opioid addiction (e.g., methadone or buprenorphine).
7. Patients with uncontrolled seizures or convulsive disorder.
8. Patients who have a confirmed diagnosis of ongoing irritable bowel syndrome.
9. Patients with evidence of clinically significant gastrointestinal disease (e.g. paralytic ileus, peritoneal carcinosis), significant structural abnormalities of the gastrointestinal tract (e.g. scarring, obstruction etc).
10. Patients who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry.
11. Surgery completed prior to the start of the study, or planned surgery during the study that would influence pain or bowel function during the study or preclude completion of the study.
12. Patients presently taking, or who have taken, naloxone <30 days prior to the start of the study.
13. Patients suffering from diarrhoea and/or opioid withdrawal.
14. Patients with any situation in which opioids are contra-indicated, severe respiratory depression with hypoxia and/or hypercapnia, severe obstructive pulmonary disease, cor pulmonale, severe bronchial asthma, paralytic ileus.
15. Patients with myxodema, hypothyroidism, Addisons disease, increase of intracranial pressure and/or epilepsy (see also exclusion criteria 7).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Patient preference of OXN compared to previous analgesics with respect to QOL
  The patient preference of OXN treatment compared to previous WHO step I or II analgesics with respect to quality of life, measured at 5 categories, as Week 2, 3, 4 of the core study (core study Week 1-4)

SECONDARY OUTCOMES:
BFI, Bowel movement, Pain relief (NAS), QOL (EQ-5D)
  The patient preference of OXN treatment compared to previous WHO step I or II analgesics with respect to overall treatment, measured at 5 categories, at Week 2, 3, 4 of the core study (core study Week 1-4). Bowel Function Index (BFI), 3 questions, at week 1-4 of the core study. Bowel movement, 2 questions, at week 1-4 of the core study. Pain relief (NAS, 0-100), at week 1-4 of the core study. Quality of Life (EQ-5D), 5 questions, at week 1 and 4 of the core study.

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels, Belgium